CLINICAL TRIAL: NCT01018485
Title: Double-Blind, Randomized, Controlled, Cross-over Comparison of Efficacy and Safety of Botulinum Toxin Type A in the Targeted Treatment of Disabling Tremor in Multiple Sclerosis
Brief Title: The Efficacy of Botulinum Toxin in Disabling Multiple Sclerosis (MS) Tremor
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Melbourne Health (Other)
Collaborators: Eastern Health (Other)
Responsible Party: Dr Andrew Evans, Royal Melbourne Hospital, Neurologist
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HREC 2008.022
Record Dates: First submitted 2009-11-19; First posted 2009-11-23 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Multiple Sclerosis; Tremor
MeSH Terms: conditions — Multiple Sclerosis; Tremor | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Botulinum Toxin First Dose (Experimental): Blinded and Randomized injection of 20 upper limbs with Botulinum Toxin Type A
  Interventions: Drug: Botulinum Toxin Type A
- Botulinum Toxin Second Dose (Experimental): 20 patients will receive Placebo as first dose and Botulinum Toxin as second dose injection 3 months after initiation of the study
  Interventions: Drug: Botulinum Toxin Type A

INTERVENTIONS:
Drug: Botulinum Toxin Type A — Intramuscular injection in affected limb up to 100 Units. Two doses (one placebo, one active) 3 months apart.
  Other Names: Botox

SUMMARY:
The incidence of tremor in Multiple Sclerosis (MS) has been estimated to affect up to 2/3rds of patients. Over half of the tremors involve the upper limb and frequently lead to further disability. Medical treatment of MS tremor is generally unrewarding, although carbamazepine, clonazepam, glutethimide, hyoscine, isoniazid, ondansetron, primidone, and tetrahydrocannabinol have been reported to have some beneficial effect but published evidence of effectiveness is very limited. The investigators' experience to date suggests that many of the upper limb tremors may potentially be responsive to Botulinum toxin injection therapy.

Aims:

1. The investigators aim to determine the efficacy of commonly used doses of BOTOX on the patients with symptomatic unilateral or bilateral arm tremor due to MS; and any side effects associated with this treatment.

ELIGIBILITY:
Inclusion Criteria:

* Relapsing-remitting MS or secondary progressive MS according to the Mc Donald criteria
* Age 18-80 years of age
* Competent to understand and sign informed consent
* Presence of symptomatic head and/or limb tremor

Exclusion Criteria:

* Treatment with botulinum toxin type A of any brand within the 4 months prior to enrollment
* A known contraindication to Botox injection
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-10; Primary Completion 2010-02 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
A decrease in tremor | 6 months

SECONDARY OUTCOMES:
The safety profile of Botulinum Toxin in MS patients | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Evans, MD, Principal Investigator — Melbourne Health
Locations (1):
- Melbourne Health, Melbourne, Victoria, Australia